CLINICAL TRIAL: NCT06549166
Title: Effectiveness of Exercise Training and Virtual Reality on Disability, Pain and Joint Position Sense in Individuals With Chronic Neck Pain: A Randomized Controlled Study
Brief Title: Virtual Reality in Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.311.IRB1.107
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
Keywords: virtual reality; exercise; neck pain
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR and exercise (Experimental): virtual reality and neck exercises
  Interventions: Other: Experimental: VR and exercise
- exercise (Sham Comparator): only neck exercise
  Interventions: Other: Sham Comparator: exercise

INTERVENTIONS:
Other: Experimental: VR and exercise — Participants will perform a 20-minute exercise program consisting of neck joint mobility exercises, neck and scapulothoracic muscle strengthening exercises, and stretching exercises. Then, for the next 20 minutes, they will engage in active neck movements using the Oculus Quest2 headset with the Ocean Rift game.
  Arms: VR and exercise
Other: Sham Comparator: exercise — The control group will perform a 40-minute same neck exercises.
  Arms: exercise

SUMMARY:
The purpose of this study is to compare the effects of virtual reality, which encourages active neck movements, in individuals with chronic neck pain, with the control group receiving only neck exercises. Participants will be randomly divided into two groups; Half of them will be given only a neck exercises program, and the other half will be given neck exercises and virtual reality.

DETAILED DESCRIPTION:
Individuals with chronic neck pain tend to have low levels of endurance in deep neck flexor muscles. Conservative treatments for neck pain, including posture education, strengthening, range of motion, motor control, flexibility, and proprioceptive training, are recommended in clinical guidelines. Virtual reality has been shown to be beneficial in the treatment of various issues related to pain in previous systematic reviews. Distracting attention is one of the mechanisms explaining the impact of virtual reality on pain. It is believed that virtual reality reduces pain perception by influencing pain pathways.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 45
* Having a history of non-traumatic neck pain persisting for more than three months
* Having a Neck Disability Index score greater than 5 points
* Not having participated in a physiotherapy program for at least 3 months
* Being able to read and write in Turkish to understand, interpret, and respond to the questionnaires

Exclusion Criteria:

* Having a surgical history in the neck region
* Having cervical spine flexion, extension, and rotation range of motion <10 degrees
* Having a history of rheumatologic, vestibular, neurological, or cardiopulmonary diseases
* Vertigo associated with neck pain
* Osteoporosis, vertebral fractures,spinal tumors
* Presence of radiculopathy or myelopathy
* Traumatic spinal cord injury
* Neck pain associated with progressive neurological deficits or loss of strength

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | 8 weeks
  Neck disability index was used to determine the pain experience and functional disability of the participants. It consists of 10 questions concern of the pain severity, ability for personal care, lifting weight, job capability headache intensity, concentration, quality of sleeping and driving and recreation activities. Total score ranges between 0 to 50 points. Zero to four points mean "no disability", 5 to 14 points mean "light disability", 15 to 24 points mean "moderate disability", 25 to 34 points mean "severe disability", and 35 to 50 points mean "complete disability".

SECONDARY OUTCOMES:
Visual analog scale | 8 weeks
  Visual analog scale is a self-reported scale consisting of a horizontal line (10 cm long) with anchor points of zero for "no pain" and ten for "worst possible pain." The patient was asked to put a mark on the line that best described the severity of his or her pain between zero and ten.
Joint position sense error | 8 weeks
  The sense of joint position error will be measured using the Cervical Range of Motion Device. The individual's head will be passively brought to 50% of the joint's range of motion, and the individual will be asked to wait for three seconds to feel the position. Then, the individual will be asked to bring their head to that position with their eyes closed. This process will be repeated three times for all directions.
Pressure pain threshold | 8 weeks
  A pressure algometer with a round tip measuring 1 cm² surface area will be used to assess pressure pain threshold. The sternum will be used as a reference point, and the trapezius and levator scapula muscles will be evaluated. The tip of the algometer probe will be applied to the skin perpendicular to it at a rate of 1 kg/cm² per second. The patient will be asked to indicate when the pressure sensation turns into pain. There will be a 30-second rest period between measurements, and bilateral evaluation will be performed, starting with the right side followed by the left side.
joint range of motion | 8 weeks
  Neck flexion, extension, right and left rotation, and right and left lateral flexion will be measured using the Cervical Range of Motion Device.
Bournemouth Neck Questionnaire | 8 weeks
  The Bournemouth Neck Questionnaire, individuals rank the following 7 dimensions of pain and function on a scale of 0 to 10: pain severity, physical disability, social disability, anxiety, depression, employment, and ability to control their pain.
Tampa Scale for Kinesiophobia | 8 weeks
  The Tampa Scale of Kinesiophobia was used to measure the kinesiophobia related to the pain. It is a scale with 17 items, and the scores range from 17 to 68. The higher the score is, the greater the kinesiophobia.
Pittsburgh Sleep Quality Index | 8 weeks
  The Pittsburgh Sleep Quality Index is a self-report assessment tool that evaluates sleep quality over a one-month period. A global score and seven component scores can be derived from the scale. The component scores are the following: Subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. Each component is scored on a scale from 0-3, with the total score ranging from 0-21; where a higher score describes poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghamkhar L, Kahlaee AH. Are Ultrasonographic Measures of Cervical Flexor Muscles Correlated With Flexion Endurance in Chronic Neck Pain and Asymptomatic Participants? Am J Phys Med Rehabil. 2017 Dec;96(12):874-880. doi: 10.1097/PHM.0000000000000778. PMID 28644248
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Tousignant M, Smeesters C, Breton AM, Breton E, Corriveau H. Criterion validity study of the cervical range of motion (CROM) device for rotational range of motion on healthy adults. J Orthop Sports Phys Ther. 2006 Apr;36(4):242-8. doi: 10.2519/jospt.2006.36.4.242. PMID 16676874
- [Background] Reddy RS, Meziat-Filho N, Ferreira AS, Tedla JS, Kandakurti PK, Kakaraparthi VN. Comparison of neck extensor muscle endurance and cervical proprioception between asymptomatic individuals and patients with chronic neck pain. J Bodyw Mov Ther. 2021 Apr;26:180-186. doi: 10.1016/j.jbmt.2020.12.040. Epub 2020 Dec 31. PMID 33992242
- [Background] Wibault J, Vaillant J, Vuillerme N, Dedering A, Peolsson A. Using the cervical range of motion (CROM) device to assess head repositioning accuracy in individuals with cervical radiculopathy in comparison to neck- healthy individuals. Man Ther. 2013 Oct;18(5):403-9. doi: 10.1016/j.math.2013.02.004. Epub 2013 Mar 7. PMID 23473752
- [Background] Clark P, Lavielle P, Martinez H. Learning from pain scales: patient perspective. J Rheumatol. 2003 Jul;30(7):1584-8. PMID 12858463
- [Background] Bolton JE, Humphreys BK. The Bournemouth Questionnaire: a short-form comprehensive outcome measure. II. Psychometric properties in neck pain patients. J Manipulative Physiol Ther. 2002 Mar-Apr;25(3):141-8. doi: 10.1067/mmt.2002.123333. PMID 11986574
- [Background] Ylinen J, Takala EP, Kautiainen H, Nykanen M, Hakkinen A, Pohjolainen T, Karppi SL, Airaksinen O. Effect of long-term neck muscle training on pressure pain threshold: a randomized controlled trial. Eur J Pain. 2005 Dec;9(6):673-81. doi: 10.1016/j.ejpain.2005.01.001. PMID 16246820
- [Background] Tejera DM, Beltran-Alacreu H, Cano-de-la-Cuerda R, Leon Hernandez JV, Martin-Pintado-Zugasti A, Calvo-Lobo C, Gil-Martinez A, Fernandez-Carnero J. Effects of Virtual Reality versus Exercise on Pain, Functional, Somatosensory and Psychosocial Outcomes in Patients with Non-specific Chronic Neck Pain: A Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Aug 16;17(16):5950. doi: 10.3390/ijerph17165950. PMID 32824394
- [Background] Hanney WJ, Kolber MJ, George SZ, Young I, Patel CK, Cleland JA. Development of a preliminary clinical prediction rule to identify patients with neck pain that may benefit from a standardized program of stretching and muscle performance exercise: a prospective cohort study. Int J Sports Phys Ther. 2013 Dec;8(6):756-76. PMID 24377062
- [Background] Peolsson A, Landen Ludvigsson M, Tigerfors AM, Peterson G. Effects of Neck-Specific Exercises Compared to Waiting List for Individuals With Chronic Whiplash-Associated Disorders: A Prospective, Randomized Controlled Study. Arch Phys Med Rehabil. 2016 Feb;97(2):189-95. doi: 10.1016/j.apmr.2015.10.087. Epub 2015 Oct 26. PMID 26514296
- [Background] Falla D, Lindstrom R, Rechter L, Boudreau S, Petzke F. Effectiveness of an 8-week exercise programme on pain and specificity of neck muscle activity in patients with chronic neck pain: a randomized controlled study. Eur J Pain. 2013 Nov;17(10):1517-28. doi: 10.1002/j.1532-2149.2013.00321.x. Epub 2013 May 6. PMID 23649799